CLINICAL TRIAL: NCT01067599
Title: Novel Determinants and Measures of Smokeless Tobacco Use: Study 2 Effects of Switching Levels of Nicotine and TSNA in Products on Smokeless Tobacco Use
Brief Title: Novel Determinants and Measures of Smokeless Tobacco Use: Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01CA141531-01 (NIH); 1R01CA141531 (NIH)
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence
Keywords: Biomarkers of tobacco exposure; Smokeless Tobacco
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low nicotine (Active Comparator): Conventional smokeless tobacco product with 1) NNN plus NNK of <2 μg/gram and nicotine levels of >5 mg/g wet weight
  Interventions: Other: Low nicotine
- Medium nicotine (Active Comparator): Conventional smokeless tobacco product with ) NNN plus NNK of <2 μg/gram and nicotine levels of 3-5 mg/g wet weight.
  Interventions: Other: Medium nicotine
- High nicotine (Active Comparator): Conventional smokeless tobacco product with NNN plus NNK of <2 μg/gram and nicotine levels of <3 mg/g wet weight
  Interventions: Other: High nicotine

INTERVENTIONS:
Other: Low nicotine — Comparison of different dosages of nicotine effect on tobacco use patterns, subjective response and biomarker levels.
  Arms: Low nicotine
Other: Medium nicotine — Comparison of different dosages of nicotine effect on tobacco use patterns, subjective response and biomarker levels.
  Arms: Medium nicotine
Other: High nicotine — Comparison of different dosages of nicotine effect on tobacco use patterns, subjective response and biomarker levels.
  Arms: High nicotine

SUMMARY:
The research project will determine the level of nicotine in ST products that will lead to the greatest reduction in toxicant exposure

DETAILED DESCRIPTION:
This is a randomized, multi-site trial determining the effects of switching smokeless tobacco (ST) users to lower toxicant ST products which vary in nicotine levels on biomarkers of exposure and patterns of use. ST users will undergo a two week baseline assessment period and then randomly assigned to one of three oral tobacco products (lower NNK plus NNN product with three different levels of nicotine) for a period of 8-weeks. Follow-up will occur at 9 and 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Using a consistent and daily amount of ST with specific nicotine and tobacco-specific nitrosamine (TSNA) levels for the past year;
2. In good physical health (no unstable medical condition);
3. Stable, good mental health (e.g., no recent unstable or untreated psychiatric diagnosis, including substance abuse, as determined by the DSM-IV criteria).

Exclusion Criteria:

1. Subjects must not be currently using other tobacco or nicotine products.
2. Female subjects cannot be pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
1. To determine if switching to ST products with reduced toxicant levels will result in reduction of biomarkers of exposure and toxicity. 2. To determine the nicotine levels of ST that would lead to the greatest reduction in tobacco toxicant exposure. | 8 weeks

SECONDARY OUTCOMES:
To determine the extent to which varying low nicotine ST products leads to compensatory tobacco use. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Hatsukami, PhD, Principal Investigator — University of Minnesota
Locations (2):
- United States (2):
  - University of Minnesota, Minneapolis, Minnesota
  - Oregon Research Institute, Eugene, Oregon